CLINICAL TRIAL: NCT01762306
Title: Efficacy for Acute Pain Alleviation of 50 mg Diclofenac 1 Hour Prior to Endometrial Sampling in Cases of Abnormal Uterine Bleeding
Brief Title: Efficacy of Diclofenac on Pain During Endometrial Sampling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIOGMVA001
Record Dates: First submitted 2012-12-11; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-09

CONDITIONS: Abnormal Uterine Bleeding Unrelated to Menstrual Cycle
MeSH Terms: interventions — Diclofenac; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Potassium (Experimental): Diclofenac Potassium 50 mg PO 1 hour prior to fractional curettage
  Interventions: Drug: Diclofenac Potassium
- Folic Acid (Placebo Comparator): Folic acid 5 mg PO 1 hour prior to fractional curettage
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Diclofenac Potassium
  Other Names: Cataflam
  Arms: Diclofenac Potassium
Drug: Folic Acid
  Arms: Folic Acid

SUMMARY:
Abnormal uterine bleeding is common in Thai women. Traditionally, because of a larger number of patients, the diagnosis of its cause is performed via fractional curettage under local anesthesia such as paracervical nerve block or intravenous meperidine.

Pain is one of a common adverse effect of this procedure and this topic should be concerned by a responsible doctor.

NSAIDs, Diclofenac Potassium in this study, is known as a drug which is effective for pain control and is as effective as coxib in acute pain management. Because of its cost, easy accessible and easy administration, Diclofenac Potassium was selected to be used in this study. Its onset of action is about 1 hour and only one dose of this drug do not cause any serious side effects.

The hypothesis of this study is that "Diclofenac Potassium has an additional effectiveness for acute pain control in patients undergoing fractional curettage under paracervical nerve block due to abnormal uterine bleeding" Double blind randomised controlled trial was performed in this study with 45 patients included in each group.

ELIGIBILITY:
Inclusion Criteria:

* Thai women at the age over 35 years old
* Presenting with abnormal uterine bleeding and have a plan of performing fractional curettage

Exclusion Criteria:

* uterine anomalies
* pregnancy
* Pelvic inflammatory disease
* Uncontrolled medical conditions
* Known cases of gynecological diseases such as gynecological malignancy, abnormal pap smear
* NSAIDs allergy
* contraindicate to NSAIDs use

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Diclofenac Potassium for additional acute pain control in patient undergoing fractional curettage under paracervical block due to abnormal uterine bleeding | 1 Year
  Effectiveness of oral 50 mg Diclofenac Potassium was measured by pain score using visual dialogue scale during operation and 30, 60, 90 and 120 minutes after procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Poomtavorn Y, Phupong V. Prospective randomized, double-blinded, placebo-controlled trial of preoperative rofecoxib for pain relief in uterine curettage. Arch Gynecol Obstet. 2005 Dec;273(2):115-8. doi: 10.1007/s00404-005-0041-y. Epub 2005 Jul 27. PMID 16047182
- [Background] Manyou B, Phupong V. Prospective randomized, double-blinded, placebo-controlled trial of preoperative etoricoxib for pain relief in uterine fractional curettage under paracervical block. Eur J Obstet Gynecol Reprod Biol. 2008 Sep;140(1):90-4. doi: 10.1016/j.ejogrb.2008.02.017. Epub 2008 Apr 8. PMID 18396369
- [Background] Macintyre PE, Walker S, Power I, Schug SA. Acute pain management: scientific evidence revisited. Br J Anaesth. 2006 Jan;96(1):1-4. doi: 10.1093/bja/aei295. No abstract available. PMID 16357114
- [Background] Buppasiri P, Tangmanowutikul S, Yoosuk W. Randomized controlled trial of mefenamic acid vs paracervical block for relief of pain for outpatient uterine curettage. J Med Assoc Thai. 2005 Jul;88(7):881-5. PMID 16241013
- [Background] Moore RA, Derry S, McQuay HJ, Wiffen PJ. Single dose oral analgesics for acute postoperative pain in adults. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008659. doi: 10.1002/14651858.CD008659.pub2. PMID 21901726
- [Background] Derry P, Derry S, Moore RA, McQuay HJ. Single dose oral diclofenac for acute postoperative pain in adults. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD004768. doi: 10.1002/14651858.CD004768.pub2. PMID 19370609
- [Background] Boonyarangkul A, Leksakulchai O. Comparison of level of pain between using manual vacuum aspiration and sharp curettage in management of abnormal uterine bleeding. J Med Assoc Thai. 2011 Dec;94 Suppl 7:S57-61. PMID 22619908
- [Background] Hinchy S, Ordman, Burrell A, Vella L, Ward L. Guidelines for the Management of Acute Pain in Adults. NHS trust; 2008.